CLINICAL TRIAL: NCT02707523
Title: Prospective Pilot Clinical Trial of Azithromycin Treatment In RSV-induced Respiratory Failure In Children
Brief Title: Prospective Pilot Clinical Trial of Azithromycin Treatment In Respiratory Syncytial Virus (RSV)- Induced Respiratory Failure In Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Michele Kong, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FWA00005960
Record Dates: First submitted 2016-02-20; First posted 2016-03-14 (Estimated); Results first posted 2020-05-27 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Respiratory Syncytial Virus
Keywords: RSV; respiratory support; ICU; Azithromycin
MeSH Terms: interventions — Azithromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participant, clinical providers and study staff are masked to the intervention. The random assignment of treatment was determined by random permutation. A statistician generated the randomization schedule and provided the randomization schedule (with randomization IDs) in an excel file to the study pharmacist in charge of dispensing the appropriate treatment.
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (Placebo Comparator): Placebo controlled (normal saline) daily for 3 days
  Interventions: Drug: Placebo
- Azithromycin (10 mg/kg) (Active Comparator): 10 mg/kg IV Azithromycin daily for 3 days
  Interventions: Drug: Azithromycin 10 mg
- Azithromycin (20 mg/kg) (Active Comparator): 20 mg/kg IV Azithromycin daily for 3 days
  Interventions: Drug: Azithromycin 20mg

INTERVENTIONS:
Drug: Azithromycin 10 mg
  Other Names: Zithromax; Z-Pak
  Arms: Azithromycin (10 mg/kg)
Drug: Azithromycin 20mg
  Other Names: Zithromax; Z-Pak
  Arms: Azithromycin (20 mg/kg)
Drug: Placebo
  Arms: Control

SUMMARY:
This randomized, double-blind, placebo-controlled phase 2 trial will be conducted at a single tertiary pediatric intensive care unit (PICU). The study will include children with RSV infection who were admitted to the pediatric intensive care unit and require respiratory support via positive pressure ventilation (invasive and noninvasive).

DETAILED DESCRIPTION:
Eligible participants include all children admitted to the PICU at Children's of Alabama with a diagnosis of RSV infection and requiring positive pressure ventilation, invasive or noninvasive, including bilevel positive airway pressure (BiPAP) or high flow nasal cannula (HFNC) oxygen (ie, >1 L/kg/min of flow, with 5 L/min flow for children weighing <5 kg). During hospitalization, all patients will be treated according to the American Academy of Pediatrics guidelines for the management of bronchiolitis, primarily supportive care. Participants will then be randomized according to a permuted-block design to receive either placebo (saline) or AZM (Fresenius Kabi) at 10mg/kg/d (ie, standard dose) or 20mg/kg/d (ie, high dose) intravenously every 24 hours for 3 days. All biologic samples collected will be analyzed in the PI's lab at the University of Alabama at Birmingham. Drug pharmacokinetics will be performed at the Pharmaceutical Sciences Research Institute of Samford University, Birmingham, AL.

ELIGIBILITY:
Inclusion Criteria:

* Admission to the PICU with RSV infection
* Need for positive pressure ventilation (invasive and non-invasive)
* Randomization and drug/placebo initiation within 48 hours of admission to Pediatric Intensive Care Unit

Exclusion Criteria:

* Azithromycin use within 7 days of PICU admission
* Contraindication to azithromycin use including:

  * Patients with electrocardiogram QT interval corrected for heart rate (Qtc) ≥ 450 ms
  * Patients with significant hepatic impairment (direct bilirubin >1.5 mg/dL)
  * Known hypersensitivity to azithromycin, erythromycin, any macrolide, or ketolide drug
  * Cardiac arrhythmia
* History of pyloric stenosis
* Immunocompromised children (any cause)
* Current use of any medication known to cause QT prolongation

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-02-06 (Actual); Study Completion 2020-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michele Kong, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Kong M, Zhang WW, Sewell K, Gorman G, Kuo HC, Aban I, Ambalavanan N, Whitley RJ. Azithromycin Treatment vs Placebo in Children With Respiratory Syncytial Virus-Induced Respiratory Failure: A Phase 2 Randomized Clinical Trial. JAMA Netw Open. 2020 Apr 1;3(4):e203482. doi: 10.1001/jamanetworkopen.2020.3482. PMID 32324238

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Azithromycin (10 mg/kg) | Azithromycin (20 mg/kg)
Started | 16 | 16 | 16
Completed | 16 | 16 | 16
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Azithromycin (10 mg/kg) | Azithromycin (20 mg/kg) | Total
Number analyzed (Participants) | 16 | 16 | 16 | 48
Age, Continuous [Mean (Standard Deviation); unit: months] | 10.8 (11) | 21.6 (29) | 20.2 (23) | 17.5 (23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 7 | 22
  Male | 9 | 8 | 9 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 2
  Not Hispanic or Latino | 16 | 15 | 15 | 46
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 5 | 2 | 12
  White | 10 | 10 | 14 | 34
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 16 | 16 | 48

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-related Adverse Events as Assessed by CTCAE v4.0
Description: To determine the safety profile of AZM at 10 mg/kg and 20 mg/kg IV X 3 days in children with RSV-induced respiratory failure
Time Frame: Baseline through Day 3
Measure: Number; unit: participants
Groups:
- Control: Placebo controlled (normal saline) daily for 3 days
  Placebo
- Azithromycin (10 mg/kg): 10 mg/kg IV Azithromycin daily for 3 days
  Azithromycin 10 mg
- Azithromycin (20 mg/kg): 20 mg/kg IV Azithromycin daily for 3 days
  Azithromycin 20mg
Arm/Group | Control | Azithromycin (10 mg/kg) | Azithromycin (20 mg/kg)
Number analyzed (Participants) | 16 | 16 | 16
participants | 0 | 0 | 0

2. Primary Outcome: Nasal Total Matrix Metalloproteinase (MMP)-9 Level
Description: To determine the concentration of total MMP-9 levels in the nasal compartment
Time Frame: Day 3
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Control | Azithromycin (10 mg/kg) | Azithromycin (20 mg/kg)
Number analyzed (Participants) | 16 | 16 | 16
ng/ml | 545 (708) | 267 (301) | 413 (814)

3. Primary Outcome: Pharmacokinetic-Plasma Half Life of AZM
Description: Measurement of AZM half life in the plasma
Time Frame: From baseline to 72 hours post treatment
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Control | Azithromycin (10 mg/kg) | Azithromycin (20 mg/kg)
Number analyzed (Participants) | 16 | 16 | 16
hours | 0 (0) | 76 (17) | 102 (33)

4. Primary Outcome: Pharmacokinetic-Lung Half Life of AZM
Description: Measurement of AZM half life in the lung
Time Frame: From baseline to 72 hours post treatment
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Control | Azithromycin (10 mg/kg) | Azithromycin (20 mg/kg)
Number analyzed (Participants) | 16 | 16 | 16
hours | 0 (0) | 78 (31) | 385 (63)

5. Secondary Outcome: Duration of Mechanical Ventilation in Days
Description: Duration of mechanical ventilation in days for enrolled subjects
Time Frame: Pre-treatment through 2 weeks
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Control | Azithromycin (10 mg/kg) | Azithromycin (20 mg/kg)
Number analyzed (Participants) | 16 | 16 | 16
Days | 4.8 (3.4) | 5.6 (5.5) | 2.6 (2.8)

6. Secondary Outcome: Duration of BiPAP in Days
Description: Duration of BiPAP in days for enrolled subjects
Time Frame: Pre-treatment through 2 weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Control | Azithromycin (10 mg/kg) | Azithromycin (20 mg/kg)
Number analyzed (Participants) | 16 | 16 | 16
days | 3.6 (13.2) | 0.4 (1.5) | 0.1 (0.3)

7. Secondary Outcome: Duration of High Flow Nasal Cannula in Days
Description: Duration of High Flow Nasal Cannula in days for enrolled subjects
Time Frame: Pre-treatment through 2 weeks
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Control | Azithromycin (10 mg/kg) | Azithromycin (20 mg/kg)
Number analyzed (Participants) | 16 | 16 | 16
Days | 3.3 (4.9) | 2.4 (2) | 2.3 (1.7)

8. Secondary Outcome: Duration of Oxygenation in Days
Description: Duration of oxygenation in days for enrolled subjects
Time Frame: Pre-treatment through 2 weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Control | Azithromycin (10 mg/kg) | Azithromycin (20 mg/kg)
Number analyzed (Participants) | 16 | 16 | 16
days | 11 (8.7) | 9.6 (5.8) | 6.6 (4)

9. Secondary Outcome: Duration of Hospitalization in Days
Description: Duration of hospitalization in days for enrolled subjects
Time Frame: Pre-treatment through 2 weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Control | Azithromycin (10 mg/kg) | Azithromycin (20 mg/kg)
Number analyzed (Participants) | 16 | 16 | 16
days | 15.8 (13.1) | 11.8 (6.5) | 9.1 (4.7)

10. Secondary Outcome: Duration of PICU Stay in Days
Description: Duration of PICU stay in days for enrolled subjects
Time Frame: Pre-treatment through 2 weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Control | Azithromycin (10 mg/kg) | Azithromycin (20 mg/kg)
Number analyzed (Participants) | 16 | 16 | 16
days | 7.7 (4.4) | 8.1 (5.8) | 5.4 (2.7)

11. Other Pre Specified Outcome: Lung Matrix Metalloproteinase (MMP) Level
Description: To determine the concentration of MMP-9 levels in the lung compartment
Time Frame: Day 3
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Control | Azithromycin (10 mg/kg) | Azithromycin (20 mg/kg)
Number analyzed (Participants) | 16 | 16 | 16
ng/ml | 13743 (23831) | 1448 (1478) | 1908 (2588)

ADVERSE EVENTS:
Time Frame: From baseline through 3 weeks (for duration of PICU stay)
Arm/Group | Control | Azithromycin (10 mg/kg) | Azithromycin (20 mg/kg)
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-10): https://cdn.clinicaltrials.gov/large-docs/23/NCT02707523/Prot_SAP_000.pdf